CLINICAL TRIAL: NCT01501669
Title: Phase III Multicenter Randomized Open-label Study of Irinotecan Plus Capecitabine Versus Capecitabine in Patients Previously Treated With Anthracycline and Taxane for HER2 Negative Metastatic Breast Cancer[PROCEED]
Brief Title: Irinotecan/Capecitabine Versus Capecitabine in Patients Treated With A/T for HER2 Negative Metastatic Breast Cancer
Acronym: PROCEED
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: Asan Medical Center (Other); Chung-Ang University (Other); Inha University Hospital (Other); Korea University Anam Hospital (Other); Samsung Medical Center (Other); Severance Hospital (Other); Seoul National University Hospital (Other); Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Jungsil Ro, Chief, Center for Clinical Trials, National Cancer Center, Korea, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-11-536
Record Dates: First submitted 2011-12-27; First posted 2011-12-29 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-07

CONDITIONS: Metastatic Breast Cancer
Keywords: irinotecan; capecitabine; metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Irinotecan; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Capecitabine alone arm (No Intervention): X arm
- Irinotecan plus capecitabine arm (Experimental)
  Interventions: Drug: Irinotecan, Capecitabine

INTERVENTIONS:
Drug: Irinotecan, Capecitabine — Irinotecan 80 mg/m2, day 1 and 8, every 3 weeks
  + capecitabine 1000 mg/m2, BID, day 1-14, every 3 weeks
  Other Names: IX arm
  Arms: Irinotecan plus capecitabine arm

SUMMARY:
This study is a multicenter, randomized study, open-label, phase III study.The efficacy of irinotecan and capecitabine combination will be superior to capecitabine alone in term of progression free survival in metastatic breast cancer patients previously treated with anthracycline and taxane.

DETAILED DESCRIPTION:
Prior to enrollment, patients will be confirmed for hormone and HER2 receptor status. Patients may have either measurable and/or evaluable metastatic lesions which are able to be assessed by chest, abdomen CT and bone scan performed within 28 days prior to start of treatment.

* Capecitabine alone arm: 1250 mg/m2, BID, day 1-14, every 3 weeks
* Irinotecan plus capecitabine arm : Irinotecan 80 mg/m2, day 1 and 8, every 3 weeks + capecitabine 1000 mg/m2, BID, day 1-14, every 3 weeks.

Randomization will be done using a random block size permutation method and stratified based on : hormone receptor status (negative vs. positive), first line vs. more than second lines, visceral metastasis (negative vs. positive).

Treatment will continue until disease progression, death, or discontinuation due to side effects of drugs or refusal by patients.

The primary objective of this study is to estimate the PFS of capecitabine and irinotecan in patients with anthracycline and taxane- pretreated metastatic breast cancer, which will be estimated by the Kaplan-Meier method and compared by log-rank test. Overall survival will be also estimated by same method. The secondary statistical analysis consisting of an estimation of the complete and partial response rates and response rates of the treatment will be calculated as the ratio of the number of complete and partial responders to the total number of evaluable patients and toxicity profile, which will be estimated as the ratio of the number of occurrence to the total number of evaluable patients. A 95% confidence interval for the response rate is computed based on the binomial distribution function. The analysis for reporting the final treatment results will be undertaken when each patient has been potentially followed for a minimum of 12 months. The overall survival and progression free survival, and their respective medians will be estimated with 95% confidence intervals.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed stage IV or recurrent breast cancer
* HER2 negative disease, or HER2 unknown disease not eligible for anti-HER2 therapy
* ECOG performance status 0-2
* Age ≥ 20 years
* Patients who received anthracycline based chemotherapy in the (neo)adjuvant or metastatic setting and experienced disease progression on taxane based chemotherapy in the metastatic setting, or patients who experienced disease recurrence within 1 year after completion of (neo)adjuvant anthracycline and taxane based chemotherapy
* In case of patients treated with capecitabine in an adjuvant setting, disease recurrence should not be occurred within 1 year after completion of capecitabine chemotherapy
* Patients with brain metastasis can be enrolled when they don't need any treatment regarding to brain metastasis
* Previous any chemotherapy and radiotherapy should be completed at least 3 weeks before randomization- Measurable or evaluable disease according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 [21]
* Adequate hematopoietic function: absolute granulocyte count ≥ 1,500/mm3, platelet ≥ 100,000/mm3, hemoglobin ≥ 10g/mm3
* Adequate hepatic function: total bilirubin ≤ 1.5mg/dL, alkaline phosphatase(ALP) ≤ 2.5 x UNL, AST/ALT ≤ 2x UNL, or if liver function abnormalities due to underlying malignancy exists, AST/ALT ≤ 2.5 x UNL, total bilirubin ≤ 3.0mg/dL, (ALP) ≤ 5 x UNL in cases with bone metastasis; ALP ≤ 5 x UNL
* Adequate renal function : serum creatinine ≤ 1.5mg/dL
* Ability to understand and comply with protocol during study period
* Patients should sign a written informed consent before study entry

Exclusion Criteria:

* Pregnant or lactating women
* Patients who receive irinotecan or capecitabine for metastatic breast cancer treatment
* Patients with HER2 positive breast cancer
* Grade 2 or greater peripheral neuropathy
* Patients with symptomatic brain metastasis
* Prior unanticipated severe reaction to fluropyrimidine therapy or known sensitivity to 5-fluorouracil
* Patients who have history of cancer other than in situ cervical cancer or non-melanotic skin cancer
* Patients with GI tract disease resulting in an inability to take oral medication, malabsorption syndrome, a requirement for IV alimentation, prior surgical procedure affecting absorption, uncontrolled GI disease (e.g. Crohn's disease, ulcerative colitis)

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Estimated)
Dates: Start 2011-06; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | The analysis for reporting the final treatment results will be undertaken when each patient has been potentially followed for a minimum of 12 months
  Day between the date of enrollment to the date of disease progression or death

SECONDARY OUTCOMES:
Objective response rate Overall survival (OS) Toxicity Quality of life (QoL) Pharmacogenomic study of irinotecan and capecitabine | The analysis for reporting the final treatment results will be undertaken when each patient has been potentially followed for a minimum of 12 months
  Objective response rate Overall survival (OS) Toxicity Quality of life (QoL) Pharmacogenomic study of irinotecan and capecitabine

CONTACTS AND LOCATIONS:
Overall Officials: Jungsil Ro, Principal Investigator — National Cencer Center, Korea
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea